CLINICAL TRIAL: NCT05762120
Title: Effectiveness of a Weight Management Programme on Diabetes Remission in Obese Patients With Early Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Healthcare Group Polyclinics (Other Government)
Collaborators: Khoo Teck Puat Hospital (Other)
Responsible Party: Principal Investigator, Wern Ee Tang, Director, Clinical Research Unit and Information Management and Analytics, National Healthcare Group Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/00652
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual Care
- Intervention (Other): Weight Management Programme
  Interventions: Other: Weight Management Programme

INTERVENTIONS:
Other: Weight Management Programme — Weight Management Programme which consists of 4 phases:
  1. Very low calorie diet
  2. Low calorie diet
  3. Maintenance phase
  4. Continuance phase
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of a weight management programme in primary care in achieving diabetes remission in obese patients with early diabetes.

Potential participants are to attend a screening visit to determine eligibility. Eligible participants will be invited to participate in the trial within 3 months of screening visit. 120 participants will be recruited into the study and randomised into 2 arms: control group (60 participants) or intervention group (60 participants).

Control group: Participants randomised to the control group will receive usual care with their healthcare team.

Intervention group: Participants randomised to the intervention group will be put on a weight management programme with the aim of achieving weight loss of at least 15% body weight or 15kg.

Researchers will compare between control and intervention groups to see if a weight management programme is effective in achieving diabetes remission in obese patients with early diabetes, compared to usual care.

DETAILED DESCRIPTION:
CONTROL GROUP

Participants randomised to the control group will receive usual care that does not include very low calorie diet (VLCD). They will be offered up to 6 dietitian consultations and 6 nurse diabetes counselling sessions (optional) over 18 months (78 weeks). They will be provided a wearable device to monitor their physical activity.

INTERVENTION GROUP

Phase A - Very low calorie diet (VLCD) phase (800kcal/day) (12 weeks)

* A commercially available micronutrient-replete 840kj/201kcal liquid formula diet (shakes) will be provided (Optifast, Nestle Health Science) to replace usual foods, with ample fluids for 12 weeks.
* Soluble fibre supplements (Fybogel 2 x 3.5 g/day) will be provided to participants to reduce constipation.
* Oral hypoglycaemic agents will be withdrawn at the start of this phase. Oral hypoglycaemic agents may be reintroduced if blood glucose levels are found to be persistently elevated.
* Participants who are on antihypertensive medications will have their antihypertensive medications withdrawn. Blood pressure will be closely monitored in these participants and antihypertensives reintroduced if blood pressure levels are found to be persistently elevated.
* During this phase, continuous glucose monitoring will be carried out for the first 2 weeks.
* After the first 2 weeks of this phase, participants are encouraged to monitor their glucose levels (fasting or random) using a glucometer 2 times a week.
* If they achieve BMI below 21kg/m2 or 15% body weight loss or 15kg weight loss before 12 weeks, they will be moved into the LCD phase.
* During the VLCD phase, participants will be encouraged to maintain their usual physical activities, but not increase physical activity.
* Each participant will be provided a wearable device to monitor their physical activity levels.

Phase B - Low calorie diet (LCD) phase (1,000-1,200kcal/day) (12-14 weeks)

* Participants will transit from meal replacement in the VLCD phase to taking in normal food.
* During this phase, continuous glucose monitoring will be carried out for the first 2 weeks.
* After the first 2 weeks of this phase, participants are encouraged to monitor their glucose levels (fasting or random) using a glucometer 2 times a week.
* During this phase, participants will be reviewed at 4 to 6-weekly intervals.
* During the first 4 weeks of this phase, participants will be encouraged to maintain their usual physical activities but not increase physical activity.
* After 4 weeks in this phase, incremental physical activities will be introduced to participants who are physically able, with the aim of achieving 7,500-10,000 steps per day.
* Physical activity will be monitored using a wearable device.
* If the participants' BMI falls below 21kg/m2, or lose 15%, or 15kg of their body weight, they will be moved into the maintenance phase.

Phase C - Maintenance phase (1,200-1,500kcal/day) (24-26 weeks)

* Participants will be advised to maintain on a 1,200-1,500kcal/day food-based diet plan to support weight stabilisation and prevent weight regain.
* Participants to complete 3 day food diary before each dietitian visit.
* Continuous glucose monitoring will be carried out for the first 2 weeks of the maintenance phase.
* After the first 2 weeks of this phase, participants are encouraged to monitor their glucose levels (fasting or random) using a glucometer 2 times a week.
* Participants who are physically able will be encouraged to have regular physical activity up to a maximum of 15,000 steps per day.
* During the maintenance phase, participants will be reviewed regularly at approximately 12 to 16 weekly intervals.

Phase D - Continuance phase (24-26 weeks)

* During the continuance phase, participants will be advised to adhere to a healthy, balanced diet
* Participants to complete 3 day food diary before each dietitian visit.
* Continuous glucose monitoring will be carried out during the first 2 weeks of the continuance phase.
* After the first 2 weeks of this phase, participants are encouraged to monitor their glucose levels (fasting or random) using a glucometer 2 times a week.
* Physical activity will be monitored using a wearable device.
* Participants will be reviewed regularly at approximately 12 to 16 weekly intervals for monitoring.

METHODS AND ASSESSMENTS

* Height will be measured to the nearest mm, with the Frankfort plane horizontal, using a stadiometer.
* Body weight will be measured to the nearest 100 g in light clothing without shoes using Class 111 approved calibrated scale.
* Waist circumference will be measured halfway between the point of the lowest rib and the iliac crest.
* Hip circumference will be measured at the maximum circumference around the buttocks.
* Blood pressure will be measured with patients seated, at rest, with legs uncrossed for at least 5 minutes.
* Blood will be collected to measure electrolytes, liver function tests (ALT and AST), lipid panel, HbA1c, creatinine, fasting glucose (venous), glucose (capillary), C-peptide, urine microalbumin and full blood count.
* Physical activity will be assessed at week 12, 16, 26, 38, 52, 64 and 78 in the intervention group and at week 12, 26, 38, 52, 64 and 78 in the control group using a wearable tracker for activity and sleep tracking. The device is to be worn by participants for approximately 9 days before each data collection time point.
* Questionnaires including health-related quality of life, diabetes empowerment scale and diabetes distress scale, fat and fibre questionnaire, dietary questionnaire and physical activity questionnaire will be administered at baseline, week 26, 52 and 78 for all participants.

CONTRACEPTION AND PREGNANCY TESTING

Urine pregnancy test is performed at screening visit for women with reproductive capacity (pre-menopause without hysterectomy) to exclude pregnancy. Those who are considering pregnancy during the study period will be excluded. Women with reproductive capacity will be advised not to plan for pregnancy during the study period. Urine pregnancy test will be done at baseline, 6, 12 and 18 months (week 0, 26, 52 and 78) for all female participants with reproductive capacity. Participants who have a positive urine pregnancy test will be dropped from the study.

RELAPSE MANAGEMENT FOR WEIGHT REGAIN

If weight regain occurs, or if diabetes is found to have returned (HbA1c ≥6.5%) at any time during the first 52 week period, 'rescue plans' to reverse weight gain will be offered.

1. Weight regain of >2 kg: offer LCD using meal replacement to replace one or two main-meal per day for 4 weeks.
2. Weight gain of >4 kg, or to <15 kg below starting weight or if diabetes recurs: offer 4 weeks VLCD using meal replacement with fortnightly dietitian review and then a 2-4 weeks LCD. Individualised dietary advice and physical activity targets will be reinforced for weight loss maintenance.

EXPECTED RISKS

Expected risks to the subjects in the intervention arm are:

* when in the very low calorie diet phase of the study are symptoms of ketosis (such as feeling thirstier than usual, muscle cramps, headaches, fatigue and weakness), feeling hungry, constipation and diarrhoea.
* fluctuations in blood glucose and blood pressure

Patients will be monitored closely and medical attention given to patient when any of the symptoms are detected.

AE REPORTING AND FOLLOW-UP

Subjects will be monitored for any adverse events at each study visit. Any adverse event will be reported to the PI and followed up as appropriate.

SAE REPORTING

SAEs that are unanticipated, serious, and possibly related to the study intervention will be reported to the Independent Monitor and DSRB in accordance with requirements.

* Unexpected fatal or life-threatening AEs related to the intervention will be reported to the DSRB within 7 days. Other serious and unexpected AEs related to the intervention will be reported to the DSRB within 15 days.
* Anticipated or unrelated SAEs will be handled in a less urgent manner but will be reported to the Independent Monitor and NHG DSRB. In the annual AE summary, the Independent Monitor Report will state that they have reviewed all AE reports.

SAFETY REVIEW PLAN

Study progress and safety will be reviewed quarterly (and more frequently if needed). Progress reports, including patient recruitment, retention/attrition, and AEs, will be provided to the Independent Monitor following each of the quarterly reviews.

DESIGNATION OF AN INDEPENDENT MONITOR

The Independent Monitor for this study has been appointed from National Healthcare Group Polyclinics. The Independent Monitor is not a member of the study team and works independently of the PI.

DATA QUALITY ASSURANCE

Description of Plan for Data Quality and Management

The PI or study team member will review all data collection forms on an ongoing basis for data completeness and accuracy as well as protocol compliance.

Collected data will be verified by checking primary and secondary endpoint data against original source documents. Data verification will be performed by someone other than the individual who originally collected the data.

DATA ENTRY AND STORAGE

For hardcopy data, they will be stored in designated locked cabinet(s) or room(s) that are accessible to authorized study personnel only. For electronic data, they will be stored on in a secured computer that is password protected. The databases will not contain subject identifiers and the data linking subject identifiers and the subject identification codes will be stored separately.

SAMPLE SIZE AND STATISTICAL METHODS

Determination of Sample Size

120 participants (60 per arm) will be recruited to the study. Power calculation has assumed diabetes remission in 27% of intervention participants at one year compared with 5% in the control group. Recruitment of at least 42 participants per arm will provide over 80% power at alpha = 0.05. Allowing for an estimated 30% individual participant drop-out within 12 months (52 weeks), we will recruit a total of 120 participants (60 per arm).

Statistical and Analytical Plans

Primary outcome measures will be analysed in a hierarchical fashion, first analysing reduction in weight of 15% body weight or 15 kg or more as a binary outcome with significance assessed at the 5% significance level, followed, if the first test is significant, by test of remission of diabetes status as a binary outcome also at the 5% level of significance. Outcome data will be analysed initially on an intention-to-treat (ITT) basis at the 18 months (78 weeks) time point. Participants reporting drug intolerance, diet intolerance or poor-compliance will be recorded and these participants will be included in the ITT analysis. For participants who discontinue the formal weight management programme the best available follow-up weights and the end of study diabetes status will be used.

Descriptive analyses will be obtained for patients in both groups. Continuous variables will be presented as mean (SD) or median (range) while categorical variables will be reported as frequencies and percentages. Plots will be generated to highlight the distribution of observations or trends. Based on the normality distribution of continuous data, the test for significance will be performed using either independent t-test or Mann-Whitney U test as appropriate. Dichotomous and categorical data will be performed using the Fisher's exact test. A p-value of < 0.05 will be regarded as statistically significant. A secondary per protocol 'completer's analyses' of those who complete the intended management will be performed as well. Data will be analysed using Stata version 17.0 for Windows (StataCorp LLC, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* Singaporean citizen or Singaporean Permanent Resident
* Age between 21 to 60 years old
* BMI between 27 to 45kg/m2
* Type 2 Diabetes Mellitus diagnosis of less than 5 years duration
* Recent HbA1c more than or equals to 6.5% if patient is on diet management alone
* Recent HbA1c more than or equals to 6.1% if patient is on treatment with oral hypoglycaemic agents
* Able to consume food products containing fish oil
* Able to consume dairy products
* Able to commit to study duration

Exclusion Criteria:

* Current insulin use
* Current treatment with anti-obesity drugs
* Recent HbA1c more than or equals to 12%
* Recent eGFR < 60 mL/min/1.73m2
* History of diabetic retinopathy
* History of ischaemic heart disease, myocardial infarction or cardiac failure
* History of cerebrovascular event
* Known liver cirrhosis
* Known cancer not in remission
* Active gout
* Active gallstone disease or known asymptomatic gallstones
* History of diagnosed eating disorder
* History of hospitalisation for depression or on antidepressants within the past 6 months
* Significant previously diagnosed psychiatric disorder eg schizophrenia, obsessive compulsive disorder
* History of substance abuse, including alcohol use disorder
* Women who are pregnant, or are considering pregnancy within the following 18 months
* Women who are breastfeeding, or are considering breastfeeding within the following 18 months
* Current participation in another research trial

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Diabetes Remission | 12 months (52 weeks)
  Percentage of participants achieving HbA1c <6.5% without medications
Weight Loss | 12 months (52 weeks)
  Percentage of participants achieving weight loss of 15% or 15kg or more

CONTACTS AND LOCATIONS:
Overall Officials: Wern Ee Tang, Principal Investigator — National Healthcare Group Polyclinics
Locations (1):
- National Healthcare Group Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No